CLINICAL TRIAL: NCT00203294
Title: Comparison Of Greater Occipital Nerve Block With Lidocaine And Bupivicaine Alone Or With Steroids In a Chronic Headache Population
Brief Title: A Research Study to Examine the Difference Between Local Anesthetics Alone and Local Anesthetics Plus Steroids in the Treatment of Chronic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GONB/ STE/ 01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Lidocaine; Sodium Chloride; Triamcinolone; Steroids; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine 2%, Bupivicaine 0.5% and saline (Active Comparator): Adult patients with CDH, and headache of at least moderate intensity at time of treatment, were randomized to receive bilateral GONB and trigger point injections in the cervical paraspinal and the trapezius muscles bilaterally.
  Interventions: Drug: lidocaine, bupivicaine and saline
- Lidocaine 2%, Bupivicaine 0.5% and triamcinolone 40 mg (Active Comparator): Adult patients with CDH, and headache of at least moderate intensity at time of treatment, were randomized to receive bilateral GONB and trigger point injections in the cervical paraspinal and the trapezius muscles bilaterally.
  Interventions: Drug: lidocaine plus bupivicaine plus triamcinolone (steroid)

INTERVENTIONS:
Drug: lidocaine, bupivicaine and saline — lidocaine, bupivicaine and saline-2 cc were injected to each GON and 0.5 cc to each trigger point. Total injected volume = 10 cc.
  Arms: Lidocaine 2%, Bupivicaine 0.5% and saline
Drug: lidocaine plus bupivicaine plus triamcinolone (steroid) — lidocaine, bupivicaine and triamcinolone (steroid)-2 cc were injected to each GON and 0.5 cc to each trigger point. Total injected volume = 10 cc.
  Other Names: Kenalog
  Arms: Lidocaine 2%, Bupivicaine 0.5% and triamcinolone 40 mg

SUMMARY:
Subjects are scheduled to undergo a Greater Occipital Nerve Block (GONB) as treatment for your chronic daily headache (CDH). GONB has been used for many years in the treatment of headaches. The nerve block is done by injecting a liquid drug through the skin of the back of the head to the area of the greater occipital nerve. The nerve runs superficially in this area, therefore the drugs are injected just under the skin. The injected drugs block electrical transmission through the nerve, resulting in reduced head pain. There are treatment options for patients receiving a GONB, however, some clinicians use local anesthetics (lidocaine and /or bupivicaine) alone, and some use local anesthetics with local steroid injection. The purpose of this study is to evaluate whether or not there is an observed difference between these two treatment approaches for GONB. We expect to enroll 60 patients into this research study at Thomas Jefferson University only.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 18-65 inclusive
* Patients who have chronic daily headache (15 or more headache days per month) for at least 3 months prior to enrollment in the study.
* Headache level should be 5/10 or more at time of GON block.
* Patients should have posterior cervical muscle tenderness at time of nerve block.

Exclusion Criteria:

* Patients who had surgery or any other invasive procedure in the occipital area.
* Patients with abnormal sensory findings on examination or any known neurological disease that may affect skin sensation (peripheral neuropathy, multiple sclerosis, stroke, etc).
* Patients diagnosed with cluster headache
* Patients with skin diseases that may affect skin sensation.
* Patients who are cognitively impaired.
* Patients with significant psychiatric disorder that may affect their understanding of the study protocol and/or their cooperation with the investigators.
* Patients who are pregnant or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-06; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Silberstein, MD, Principal Investigator — Thomas Jefferson University, Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- GON Block Only: Patients were injected with lidocaine 2% and bupivacaine 0.5% (in a 1:1 ratio) plus saline. Two cc were injected to each GON (greater occipital nerve) and 0.5 cc to each trigger point, to a total injected volume of 10 cc.
- GON Block Plus Steroid: Patients were injected with lidocaine 2% and bupivacaine 0.5% (in a 1:1 ratio) plus triamcinolone 40 mg. Two cc were injected to each GON and 0.5 cc to each trigger point, to a total injected volume of 10 cc.
Period: Overall Study
Arm/Group | GON Block Only | GON Block Plus Steroid
Started | 22 | 23
Completed | 14 | 10
Not Completed | 8 | 13
Not completed — Withdrawal by Subject | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GON Block Only | GON Block Plus Steroid | Total
Number analyzed (Participants) | 22 | 23 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 37
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 22 | 23 | 45

OUTCOME MEASURES:

1. Primary Outcome: Headache Severity as Measured on an 11-point Verbal Scale (0 to 10):0=No Pain 10=Excruciating Pain
Description: Headache severity was assessed on an 11-point verbal scale twenty minutes after treatment
Time Frame: 20 minutes
Population: There were 15 patients in group A (no steroids injected) and 14 in group B (steroids injected).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lidocaine 2% and Bupivacaine 0.25% Plus Saline; Lidocaine 2% and Bupivacaine 0.25% Plus Triamcinolone 40 mg.: Adult patients with Chronic Daily Headache (CDH), and headache of at least moderate intensity at time of treatment, were randomized to receive bilateral GONB and 12 trigger point injections
Arm/Group | Lidocaine 2% and Bupivacaine 0.25% Plus Saline | Lidocaine 2% and Bupivacaine 0.25% Plus Triamcinolone 40 mg.
Number analyzed (Participants) | 15 | 14
units on a scale | -3.29 (2.76) | -3.70 (1.49)
Statistical Analysis 1: Comparison: Lidocaine 2% and Bupivacaine 0.25% Plus Saline vs Lidocaine 2% and Bupivacaine 0.25% Plus Triamcinolone 40 mg; Fisher's exact test was used to compare nominal variables between groups. The Wilcoxon rank-sum test was used to compare interval and ordinal variables between groups; Test type: Superiority or Other; p < 0.01, Fisher Exact — Separate models were fit to the change scores for headache pain, nausea and vomiting, photophobia, phonophobia, and neck pain
Statistical Analysis 2: Comparison: Lidocaine 2% and Bupivacaine 0.25% Plus Saline vs Lidocaine 2% and Bupivacaine 0.25% Plus Triamcinolone 40 mg; Fisher's exact test was used to compare nominal variables between groups; Test type: Superiority or Other; p < 0.01, Fisher Exact; Wilcoxon rank-sum test was used to compare interval and ordinal variables between groups

2. Primary Outcome: Decrease in Headache Pain, as Measured on an 11-point Pain Scale (0=no Pain, 10=Excruciating Pain). Change in Headache Pain 20 Minutes After Injection Will be Compared Between Treatment Groups.
Time Frame: 20 minutes
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: pain unit

3. Secondary Outcome: To Evaluate the Effect of Treatment on Neck Pain in the Two Groups Compared to Historical Baseline, and Between the Two Treatment Groups.
Time Frame: 20 minutes
Reporting Status: Not Posted

4. Secondary Outcome: To Evaluate Effect of Treatment on Associated Symptoms (Nausea, Phonophobia and Photophobia) as Measured Using a 4 Point Scale (None, Mild, Moderate, Severe) Compared to Historical Baseline, and Between the Two Treatment Groups.
Time Frame: 20 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | GON Block Only | GON Block Plus Steroid
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23
Other Adverse Events (participants affected / at risk) | 0/22 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes